CLINICAL TRIAL: NCT07192432
Title: A Phase 1/2, First-in-Human Study of VNX-202 Gene Therapy in Patients With HER2-Positive Cancer
Brief Title: Gene Therapy for HER-Positive Cancer (SENTRY-HER2)
Acronym: SENTRY-HER2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vironexis Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VNX-202-01
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: HER2 Expressing Solid Tumors
Keywords: HER2+ breast cancer; HER2+ gastric cancer; Other HER+ cancer; HER2-low cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group 1/Group 2/Group 3/Group 4 (Experimental)
  Interventions: Genetic: Dose Level 1, VNX-202; Genetic: Dose Level 2, VNX-202; Genetic: Dose Level 3, VNX-202; Genetic: Dose Level 4, VNX-202

INTERVENTIONS:
Genetic: Dose Level 1, VNX-202 — Adeno-associated viral vector encoding the CD3/HER2 Bi-Specific T-Cell Engager (AAV.CD3/HER2), Single IV Infusion
Genetic: Dose Level 2, VNX-202 — Adeno-associated viral vector encoding the CD3/HER2 Bi-Specific T-Cell Engager (AAV.CD3/HER2), Single IV Infusion
Genetic: Dose Level 3, VNX-202 — Adeno-associated viral vector encoding the CD3/HER2 Bi-Specific T-Cell Engager (AAV.CD3/HER2), Single IV Infusion
Genetic: Dose Level 4, VNX-202 — Adeno-associated viral vector encoding the CD3/HER2 Bi-Specific T-Cell Engager (AAV.CD3/HER2), Single IV Infusion

SUMMARY:
This is a Phase 1/2, first-in-human, open-label, dose-escalating and expansion trial designed to assess the safety and efficacy of VNX-202 in patients with HER2 positive cancers.

DETAILED DESCRIPTION:
VNX-202 is an investigational adeno-associated virus (AAV) gene therapy developed to express a secreted anti-HER2/anti-CD3 scFv diabody (termed GP202). GP202 binds to human epidermal growth factor receptor 2 (HER2) on the surface of cancer cells and to cluster of differentiation (CD)3 on the surface of T cells, inducing the T cells to kill the HER2-positive cancer cells.

Following a single intravenous (IV) infusion, the vector induces the liver to continuously secrete GP202 into the bloodstream, resulting in long-term, consistent serum levels of GP202. Compared with conventionally delivered protein therapies, this gene therapy approach obviates the requirement for episodic dosing and avoids a possible reduction or loss of efficacy associated with trough levels of the protein between treatment cycles.

In this 2-part study, dose-finding data from Part 1 of the study (n=~12 patients) will be used determine the dose for Part 2 in patients. Part 1 is a dose-finding PK study in adults ≥18 years old with previously treated metastatic HER2 solid tumors designed to determine the minimal dose that achieves target PK serum levels of GP202 at steady state (8-week timepoint) without dose-limited toxicities, defined as the recommended Part 2 dose (RP2D). Participants must have histologically or cytologically confirmed HER2 positive solid tumor cancers that has progressed during or following previous anti-cancer treatment. Part 2 (n=~15) will be opened following data safety monitoring board review of Part 1 data and is designed to determine the safety and pharmacokinetics (PK) of VNX-202 at the RP2D in a broader array of subjects. Part 2 will comprise of participants with early stage HER2-positive tumors who are at risk of disease relapse and/or metastasis despite having received prior systemic and/or local treatment. Each cohort will comprise ≥5 participants (Cohort A: breast cancer; Cohort B: gastric cancer; Cohort C: all otherHER2-positive tumor types). Patients will be followed for safety and efficacy up to 5 years post VNX-202 dosing.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years of age
* Histologically or cytologically confirmed diagnosis of HER-2 positive solid tumor as defined in the protocol
* Part 1: presence of advanced or metastatic disease that has progressed during or following previous treatment
* Part 2: Early stage HER-2 positive cancers with high risk for relapse following completion of SOC or after neoadjuvant systemic treatment
* AAV specified capsid total antibody ≤1:400
* ECOG performance status of 0 or 1
* Life expectancy ≥3 months
* Protocol-specified ranges for renal, liver, cardiac and pulmonary function
* Protocol-specified ranges for hematology parameters

Exclusion Criteria:

* Hepatoxicity (AST or ALT > 2x upper limit of normal)
* Known active CNS or leptomeningeal disease
* History of thrombotic microangiopathy or cardiomyopathy, or evidence of sensory neuropathy
* Pregnant or nursing (lactating) women
* History of other malignancy within 5 years prior to screening as defined in protocol
* History of hypersensitivity to corticosteroids or history of corticosteroid-related toxicity Concurrent anti-cancer treatment in another investigational trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2033-09 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TESAEs) | Change from Baseline to Year 5 post dosing

SECONDARY OUTCOMES:
Change from baseline in T cell subsets and clonality | Change from baseline to year 5 post dosing
Change from baseline in ctDNA | Change from baseline to year 5 post dosing
Change from baseline in progression free survival | Change from baseline to year 5 post dosing
Change from baseline in overall survival | Change from baseline to year 5 post dosing

OTHER OUTCOMES:
Change in VNX-202 gene product levels | Change from baseline to year 5 post dosing
Change in VNX-202 vector shedding | Change from baseline to year 5 post dosing

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Valkyrie Clinical Trials, Los Angeles, California
  - SCRI Denver DDU at HealthOne, Denver, Colorado
  - SCRI Oncology Partners, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No